CLINICAL TRIAL: NCT07239284
Title: Efficacy and Safety of Endovenous Ablation for Relief of Knee Pain in Elderly Patients With Lower Extremity Varicose Veins: A Prospective Observational Study
Acronym: EVA-Knee-Elder
Status: Not yet recruiting | Type: Observational
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chunshui He, Ph.D , Chief Physician of Vascular Surgery , Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu University of Traditional Chinese Medicine
Other Study IDs: chengduUTCM knee-80
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Varicose Veins of Lower Limb; Chronic Venous Insufficiency, CVI; Knee Pain; Knee Osteoarthritis; Elderly Patients
MeSH Terms: conditions — Blindness, Cortical; Osteoarthritis, Knee | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endovenous Ablation for Varicose Veins — Participants will receive standard endovenous treatment for lower limb varicose veins as part of their routine clinical care. The procedure may include radiofrequency ablation (RFA), endovenous laser ablation (EVLA), or other accepted thermal ablation techniques, with or without adjunctive phlebectomy or foam sclerotherapy if clinically indicated. The intervention is performed under tumescent local anesthesia by vascular surgeons according to established guidelines. No experimental techniques or investigational devices are used.
  Other Names: Endovenous Thermal Ablation; Radiofrequency Ablation; Endovenous Laser Ablation

SUMMARY:
Lower extremity varicose veins (LEVV) are common among elderly patients and can cause leg heaviness, pain, and swelling. In some older adults, venous congestion may contribute to knee or peri-knee pain, which is often misattributed to degenerative joint disease alone. Evidence on whether varicose vein treatment can relieve knee pain in very elderly patients (aged 80 years or older) is limited.

This prospective cohort study aims to evaluate the effectiveness and safety of endovenous ablation (EVA) for improving knee pain in elderly patients with symptomatic varicose veins. The study will include participants aged 80 years or older who present with both lower extremity varicose veins and knee joint pain. Eligible patients will undergo endovenous thermal ablation (radiofrequency or endovenous laser ablation) as the primary intervention.

Participants will be assessed at baseline, 1 month, 3 months, 6 months, and 12 months after treatment. The primary outcome is the change in knee pain intensity measured by the Visual Analog Scale (VAS) from baseline to 6 months. Secondary outcomes include changes in knee joint function (assessed by the Western Ontario and McMaster Universities Osteoarthritis Index [WOMAC] or Knee Injury and Osteoarthritis Outcome Score [KOOS]), venous clinical severity score (VCSS), limb heaviness, quality of life (assessed by EQ-5D), and procedure-related complications.

Safety will be evaluated by recording peri-procedural adverse events, including deep vein thrombosis, skin burns, nerve injury, and postoperative infection. The study will also analyze whether preexisting osteoarthritis, venous reflux severity, or body mass index (BMI) affect the magnitude of pain improvement.

The hypothesis is that endovenous ablation improves knee pain in elderly patients by reducing venous congestion around the knee and improving venous return. This study will help clarify whether treating varicose veins can provide additional benefits for knee pain and mobility in patients aged 80 years and older.

ELIGIBILITY:
Inclusion Criteria:

Adults aged ≥80 years. Clinical diagnosis of lower limb varicose veins with documented venous reflux on duplex ultrasound (CEAP C2-C4).

Presence of knee pain lasting ≥4 weeks prior to enrollment, confirmed by patient-reported VAS/NRS ≥3 at baseline.

Planned to undergo standard endovenous treatment (radiofrequency ablation, endovenous laser ablation, or equivalent).

Ability to provide informed consent and complete study questionnaires.

Exclusion Criteria:

Prior surgery or endovenous ablation for varicose veins in the same limb. History of inflammatory arthritis (e.g., rheumatoid arthritis, gout) or other systemic rheumatologic disease.

Recent acute knee injury (ligament, meniscus, fracture) within 6 months. Prior knee replacement or major knee surgery. Recent intra-articular injection or arthroscopy (<3 months). Known deep vein thrombosis or history of pulmonary embolism within the past 6 months.

Severe peripheral arterial disease (ABI <0.8). Pregnancy or breastfeeding. Inability to comply with follow-up schedule or complete questionnaires.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This study will enroll elderly patients aged 80 years or older who are diagnosed with primary lower extremity varicose veins and who also experience knee or peri-knee pain. Participants will be recruited from the outpatient vascular surgery clinics and inpatient wards of the participating hospital. All participants must be ambulatory and able to complete pain and function questionnaires. The study population represents older adults who are candidates for endovenous ablation under tumescent local anesthesia and who may benefit from venous reflux correction.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-12-10 (Estimated); Study Completion 2027-07-10 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Pain Score (VAS) | Baseline, 1 month, 3 months, and 6 months
  Visual Analog Scale (VAS, 0-10 cm)
Change in Knee Function and Symptoms | Baseline, 1 month, 3 months, and 6 months
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) evaluates knee-related pain, stiffness, and functional limitations.Scoring Range: 0 to 96, with higher scores indicating worse symptoms and greater functional impairment.

SECONDARY OUTCOMES:
Change in Venous Clinical Severity Score (VCSS) | Baseline, 1 month, 3 months, and 6 months.
  The Venous Clinical Severity Score (VCSS) assesses the severity of chronic venous disease and varicose vein-related symptoms.Scoring Range: 0 to 30, with higher scores indicating more severe venous disease.
Change in Aberdeen Varicose Vein Questionnaire (AVVQ) | Baseline, 1 month, 3 months, and 6 months.
  The Aberdeen Varicose Vein Questionnaire (AVVQ) measures varicose vein-specific quality of life.Scoring Range: 0 to 100, with higher scores indicating worse quality of life.
Change in Health-Related Quality of Life | Baseline, 1 month, 3 months, and 6 months
  The Chronic Venous Insufficiency Questionnaire (CIVIQ-14) is a 14-item disease-specific instrument used to assess quality of life in patients with chronic venous disease. It covers domains of pain, physical function, and psychological impact. Scoring Range: 0 to 100, with higher scores indicating worse quality of life.
Use of Analgesic Medications | 6 months.
  Number of patients using NSAIDs or other pain medications for knee pain.
Adverse Events Related to Procedure | Within 6 months after procedure.
  Number and type of adverse events (nerve injury, phlebitis, DVT, infection).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cao TN, Nguyen CT, Nguyen MD. The association between chronic venous disease and knee osteoarthritis. Eur Rev Med Pharmacol Sci. 2023 Apr;27(7):2899-2907. doi: 10.26355/eurrev_202304_31921. PMID 37070890
- [Result] Lesnyak OM, Zubareva EV, Goncharova MG, Maksimov DM. [Lower extremity venous diseases in primary knee osteoarthritis]. Ter Arkh. 2017;89(5):53-59. doi: 10.17116/terarkh201789553-59. Russian. PMID 28631699
- [Result] Oga Y, Sugiyama S, Matsubara S, Inaki Y, Matsunaga M, Shindo A. The Effectiveness of Endovenous Thermal Ablation for the Knee Symptoms of the Osteoarthritis with Varicose Veins. Ann Vasc Dis. 2021 Jun 25;14(2):108-111. doi: 10.3400/avd.oa.21-00016. PMID 34239634
- [Result] Gunes S, Sehim K, Cuneyt K, Gokmen D, Kucukdeveci AA. Is there a relationship between venous insufficiency and knee osteoarthritis? Turk J Phys Med Rehabil. 2020 Mar 3;66(1):40-46. doi: 10.5606/tftrd.2020.5110. eCollection 2020 Mar. PMID 32318673